CLINICAL TRIAL: NCT02570243
Title: High (100IU/Kg) Versus Standard (50IU/Kg) Heparin Dose for Prevention of Forearm Artery Occlusion Forearm Artery Occlusion
Brief Title: High (100IU/Kg) Versus Standard (50IU/Kg) Heparin Dose for Prevention of Forearm Artery Occlusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor of Cardiology, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY 20
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Coronary Angiography
Keywords: heparin; radial artery
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard dose of Heparin (Active Comparator): 50IU/Kg heparin intravenously
  Interventions: Drug: Standard dose of Unfractionated heparin
- High dose of Heparin (Experimental): 100IU/Kg heparin intravenously
  Interventions: Drug: High dose of Unfractionated Heparin

INTERVENTIONS:
Drug: High dose of Unfractionated Heparin — Unfractionated Heparin 100IU/Kg
  Arms: High dose of Heparin
Drug: Standard dose of Unfractionated heparin — Unfractionated heparin 50IU/Kg
  Arms: Standard dose of Heparin

SUMMARY:
This is a prospective, multi-center, superiority study of parallel design. Patients are enrolled if they are older than 18 years old, are scheduled for 5 or 6 Fr diagnostic coronary angiography and the interventional cardiologist is willing to proceed with radial access. Patients are randomized before diagnostic catheterization to receive intravenously either 100IU/Kg or 50 IU/Kg of unfractionated heparin (UFH) in a 1:1 ratio. Patients are discharged usually within 4 to 6 hours after coronary angiography.

Radial artery in each patient is evaluated either in-hospital or during a subsequent visit by one physician who is blinded to the actual antithrombotic treatment given. Radial artery is considered occluded if it exhibits ultrasonographically no antegrade flow signal both at baseline and after reevaluation on a second occasion, within 30 days after the index procedure. Initially patent arteries will not be reexamined and are thought to remain permanently patent. The investigators also monitor major bleeding (defined as ≥ 5g/dL decrease in hemoglobin or ≥15% decrease in hematocrit or any life-threatening bleeding (confirmed by MRI or computed tomography) and large local hematomas of the forearm (defined as those extending beyond the forearm).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Scheduled for 5 or 6 Fr diagnostic coronary angiography
* The interventional cardiologist is willing to proceed with radial access
* Written informed consent

Exclusion Criteria:

Before randomization

* chronic hemodialysis
* oral anticoagulation
* hemodynamic instability
* severe dermo-myoskeletal forearm deformities
* history of CABG and bilateral use of either the internal mammary or radial artery
* history of CABG and ipsilateral use of both the internal mammary and radial artery
* admission for elective PCI After randomization
* crossover to another arterial access site is required
* ad hoc PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2015-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Radial artery occlusion | 30 days
  Radial artery occlusion as assessed by Doppler Ultrasound

SECONDARY OUTCOMES:
Large local hematomas of the forearm | 30 days
  large local hematomas of the forearm (defined as those extending beyond the forearm)
Major bleeding | 30 days
  ≥ 5g/dL decrease in hemoglobin or ≥15% decrease in hematocrit or any life-threatening bleeding (confirmed by MRI or computed tomography)

CONTACTS AND LOCATIONS:
Locations (1):
- Patras University Hospital, Pátrai, Rion, Greece

REFERENCES:
- [Derived] Hahalis GN, Leopoulou M, Tsigkas G, Xanthopoulou I, Patsilinakos S, Patsourakos NG, Ziakas A, Kafkas N, Koutouzis M, Tsiafoutis I, Athanasiadis I, Koniari I, Almpanis G, Anastasopoulou M, Despotopoulos S, Kounis N, Dapergola A, Aznaouridis K, Davlouros P. Multicenter Randomized Evaluation of High Versus Standard Heparin Dose on Incident Radial Arterial Occlusion After Transradial Coronary Angiography: The SPIRIT OF ARTEMIS Study. JACC Cardiovasc Interv. 2018 Nov 26;11(22):2241-2250. doi: 10.1016/j.jcin.2018.08.009. Epub 2018 Nov 1. PMID 30391389